CLINICAL TRIAL: NCT06532474
Title: Pilot Study Exploring the Physiologic, Pharmacodynamic, and Clinical Responses of Skeletal Muscle in Patients With Spinal Muscular Atrophy Treated With SMN-Directed Therapies
Brief Title: Exploring the Physiologic, Pharmacodynamic, and Clinical Responses of Skeletal Muscle in Patients With Spinal Muscular Atrophy Treated With SMN-Directed Therapies
Status: Recruiting | Type: Observational
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: ML43225
Record Dates: First submitted 2024-07-29; First posted 2024-08-01 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-11

CONDITIONS: Spinal Muscular Atrophy
Keywords: Spinal Muscular Atrophy (SMA); SMA drugs; Responses of Skeletal Muscle; SMN-directed therapies; Eyrysdi; Spinraza; Zolgensma
MeSH Terms: conditions — Muscular Atrophy, Spinal

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood and urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Cohort 1: Current Evrysdi prescription
- Cohort 2: Current Spinraza or Zolgensma prescription
- Cohort 3: Changing from Spinraza or Zolgensma to Evrysdi
- Cohort 4: Have never received any SMN-directed therapies

SUMMARY:
In this observational study, researchers are looking at the effects of spinal muscular atrophy (SMA) drugs on the muscles and nerve cells in patients with SMA.

Primary Objectives

* To evaluate the feasibility and reliability of performing MR functional imaging in exercising muscle in patients with SMA.
* To evaluate patients with SMA types 2 and 3 at baseline and longitudinally at 6 and 12 months

Secondary Objectives

* To describe the MR functional bioenergetics response in the leg muscles in four potential groups of patients with spinal muscular atrophy: untreated, actively treated with nusinersen (Spinraza®) or onasemnogene abeparvovec (Zolgensma®), actively treated with risdiplam (Evrysdi®), and switching from Spinraza or Zolgensma to Evrysdi.
* To identify changes in motor function in patients with SMA types 2 and 3 who initiate treatment with risdiplam.
* To obtain biomarkers in blood, urine, and muscle tissue to provide proof-of-concept support for risdiplam effect on skeletal muscle.
* To obtain quality of life and disability data from participants in this study.

DETAILED DESCRIPTION:
This is an observational study to demonstrate the feasibility of performing MR functional imaging in exercising muscle in patients with SMA. The participants will be prescribed medication by their treating physician, they will not receive any drug as part of this study.

Participants participating in the ML43225 study, will be put into one of four groups depending on their type of SMA and the drugs they may or may not be taking. They will be asked to come to clinic 3 times over one year. Each visit will include magnetic resonance (MR) studies, a muscle ultrasound, a nerve test, muscle function testing, lung function testing, blood work, vital signs, and participants will be asked about their quality of life and daily life activities. After participants have completed the 3 required visits, they will be taken off study.

ELIGIBILITY:
Inclusion Criteria:

* Genetic confirmation of SMA with homozygous deletion of SMN1 or compound heterozygous deletion/mutation of SMN1
* Two, three, or four copies of SMN2
* Age 5 to 20 years
* Non-ambulatory participants: maximum function sitting or standing with support, never walked independently, still able to sit independently for 5 seconds at screening, with active ankle plantar flexion strength of at least 3 N with hand-held myometry and capable of performing repetitive maximal plantar flexion effort for 120 seconds. HFMSE score at screening between 10 and 45 points.
* Ambulatory participants: minimum function of independent walking, able to walk unassisted a minimum of 100 meters at screening, ankle plantar flexion strength of at least 10 N with hand-held myometry and capable of performing repetitive maximal plantar flexion for 120 seconds. HFMSE score at screening between 40 and 60.
* SMN-directed therapy inclusion:

  * Current Evrysdi prescription

    * Must have Evrysdi prescription through their treating physician but have not yet initiated treatment OR
  * Current Spinraza or Zolgensma prescription

    * For patients on Spinraza, must have been taking Spinraza for at least 12 months at screening (4 loading and 2 maintenance doses) and following the FDA-recommended dosing schedule
    * For patients on Zolgensma, must have been dosed at least one year prior to screening
    * Must have Spinraza or Zolgensma prescription through their treating physician OR
  * Changing from Spinraza or Zolgensma to Evrysdi

    * For patients on Spinraza, must have been taking Spinraza for at least 12 months at screening (4 loading and 2 maintenance doses) and following the FDA-recommended dosing schedule
    * For patients on Zolgensma, must have been dosed at least one year prior to screening
    * Must have voluntarily decided to switch therapies based on discussion with their treating physician
    * Must have Evrysdi prescription through their treating physician but have not yet initiated treatment OR
  * Have never received any SMN-directed therapies

Exclusion Criteria:

* Labs at screening that are abnormal and identified as clinically significant by the PI: CBC, and CMP, liver function tests (over twice the upper limit of normal), PT/PTT, urine protein of 2+ or greater.
* Inability to perform reliably the motor function testing or the exercise testing in the MR scanner.
* Treatment with a possible SMA-enhancing or mitochondrial-enhancing medication, unless discontinued within 3 months prior to screening: oral albuterol, hydroxyurea, phenylbutryate, valproic acid, creatine, l-carnitine, or other mitochondrial type supplement (riboflavin, lipoic acid, etc.). A daily multivitamin and Vitamin D supplement and intermittent inhaled albuterol are permitted if the dosage is unchanged during the study.
* Need for routine non-invasive ventilation support.
* Non-oral nutritional support, e.g., gastrostomy tube feeding.
* Any ferrous metal implants (e.g., spinal rods) that preclude testing in a MR scanner.

Ages: 5 Years to 20 Years | Sex: All
Age Groups: Child, Adult
Study Population: Those who meet the Eligibility criteria and consent to enrollment on the study.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2025-10-29 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Feasibility of performing MR functional imaging in SMA patients | At baseline and at 6 months (+/- 14 days)
  MR functional imaging is considered feasible if ≥ 80% of MRI protocol eligible patients can complete 100% of imaging assessments at baseline and 6 months.
Reliability of performing MR functional imaging in SMA patients | At baseline and at 6 months (+/- 14 days)
  MR functional imaging is considered reliable if the test-retest reliability is ≥ 0.80 for key imaging biomarkers.
Compare skeletal muscle oxidative phosphorylation bioenergetics in patients with SMA types 2 and 3 (phosphocreatine) | At baseline and longitudinally at 6 (+/- 14 days) and 12 months (+/- 14 days)
  Real-time 31P MR spectroscopy and CrCEST MRI will be used to measure phosphocreatine within the gastrocnemius-soleus leg muscles at rest, during an exercise protocol, and during post-exercise recovery to baseline. Both measure the recovery time in seconds.
Compare skeletal muscle oxidative phosphorylation bioenergetics in patients with SMA types 2 and 3 (creatine concentrations) | At baseline and longitudinally at 6 (+/- 14 days) and 12 months (+/- 14 days)
  Real-time 31P MR spectroscopy and CrCEST MRI will be used to measure creatine concentrations within the gastrocnemius-soleus leg muscles at rest, during an exercise protocol, and during post-exercise recovery to baseline. Both measure the recovery time in seconds.
Measure intramuscular fat fraction in major muscle groups of the lower extremity in patients with SMA types 2 and 3 | At baseline and longitudinally at 6 (+/- 14 days) and 12 months (+/- 14 days)
  Measurement of thickness of muscle compared to fat on MRI, measured in percentage.
Measure electrophysiological tests of motor neuron function to repetitive nerve stimulation in patients with SMA types 2 and 3 | At baseline and longitudinally at 6 (+/- 14 days) and 12 months (+/- 14 days)
  Electrophysiological testing: Compound motor action potential (CMAP, measured in millivolts), motor unit number estimate (MUNE, average 200-400 for most limb muscles), and repetitive stimulation at 3 Hz - right ulnar to abductor digiti minimus and right fibular/peroneal nerve to tibialis anterior muscle.
  A decrease of more than 40% in the amplitude of CMAP is considered abnormal.

SECONDARY OUTCOMES:
Identify changes in motor function in non-ambulant patients and ambulant patients with SMA types 2 and 3 | At baseline and longitudinally at 6 (+/- 14 days) and 12 months (+/- 14 days)
  The Hammersmith Functional Motor Scale Expanded (HFMSE) has a score range from 0-66 with lower scores indicating poorer overall motor function.
Identify changes in motor function in non-ambulant patients with SMA types 2 and 3 - Revised Upper Limb Module | At baseline and longitudinally at 6 (+/- 14 days) and 12 months (+/- 14 days)
  The Revised Upper Limb Module (RULM) has a score range 0-37 with lower scores indicating poorer upper limb motor function.
Identify changes in motor function in non-ambulant patients with SMA types 2 and 3 - Block and Box Test | At baseline and longitudinally at 6 (+/- 14 days) and 12 months (+/- 14 days)
  The Block and Box Test (BBT) is a measure of gross manual dexterity and is scored by counting the number of blocks carried from one compartment to another. Higher scores are indicative of better manual dexterity.
Identify changes in motor function in ambulant patients with SMA types 2 and 3 - 6-Minute Walk | At baseline and longitudinally at 6 (+/- 14 days) and 12 months (+/- 14 days)
  The 6-Minute Walk (6MW) Test measures how far someone can walk in six minutes, a higher score indicates better exercise tolerance score. A low score correlates with lower function.
Identify changes in motor function in ambulant patients with SMA types 2 and 3 - 10 Meter Walk/Run | At baseline and longitudinally at 6 (+/- 14 days) and 12 months (+/- 14 days)
  The 10 Meter Walk/Run (10MW) Test is measured in seconds and assesses walking speed over a short distance. Longer times indicate lower motor function
Identify changes in motor function in ambulant patients with SMA types 2 and 3 - 4-Stair Climb | At baseline and longitudinally at 6 (+/- 14 days) and 12 months (+/- 14 days)
  The 4-Stair Climb (4SC) Test is measured in seconds and assesses lower extremity power and motor function. Longer times indicate lower motor function
Identify changes in motor function in ambulant patients with SMA types 2 and 3 - Supine-to-Stand Test | At baseline and longitudinally at 6 (+/- 14 days) and 12 months (+/- 14 days)
  The Supine-to-Stand (STS) Test is measured in seconds and assesses the ability to move from laying on your back to standing up straight. Longer times indicate lower motor function.
Identify changes in motor function in ambulant patients with SMA types 2 and 3 - Timed Up-and-Go Test | At baseline and longitudinally at 6 (+/- 14 days) and 12 months (+/- 14 days)
  The Timed Up-and-Go (TUG) Test is measured in seconds and assesses the ability to stand up from sitting in a chair, walk 10 feet, turn around, walk back, and sit down. Longer times indicate lower motor function
Assess myometry, or measurement of muscle strength | At baseline and longitudinally at 6 (+/- 14 days) and 12 months (+/- 14 days)
  Myometry measures force in pounds or kilograms and measures the strength of a muscle group. The more force measured indicates more muscle strength.
Muscle ultrasound thickness and echogenicity of 5 muscles - 2 upper limb and 3 lower limb | At baseline and longitudinally at 6 (+/- 14 days) and 12 months (+/- 14 days)
  Muscle thickness is measured in centimeters and echogenicity is measured in gray-scale value. Muscle thickness and echogenicity are related to muscle strength, physical function, muscle mass, and quality of muscle.
Plasma neurofilament light (NF-L) and phosphorylated heavy chain (pNF-H) levels | At baseline and longitudinally at 6 (+/- 14 days) and 12 months (+/- 14 days)
  The NF-L and pNF-H levels are measured in nanograms per milliliter from blood samples and can be an indicator of nerve cell damage. Higher values normally mean more nerve damage is occurring.
Blood SMN protein levels | At baseline and longitudinally at 6 (+/- 14 days) and 12 months (+/- 14 days)
  SMN protein levels are measured in nanograms per milliliter from blood samples. Higher values indicate more SMN protein production which is normally deficit in people with SMA.
Pyruvic acid (mg/dL) | At baseline and longitudinally at 6 (+/- 14 days) and 12 months (+/- 14 days)
  This parameters has been added to better understand systemic glycolysis in this population in the context of measuring bioenergetics in muscle via fMRS. A normal blood pyruvic acid level is between 0.3 and 1.5 milligrams per deciliter (mg/dL). Elevated pyruvic acid in glycolysis usually indicates a disruption in the normal metabolic pathway.
Lactic Acid (millimoles per liter) | At baseline and longitudinally at 6 (+/- 14 days) and 12 months (+/- 14 days)
  This parameter has been added to better understand systemic glycolysis in this population in the context of measuring bioenergetics in muscle via fMRS. Normally, blood lactate levels are between 1-2 mmol/L when not exercising. Elevated lactic acid during glycolysis indicates that the body is primarily relying on anaerobic glycolysis, meaning it is breaking down glucose for energy without sufficient oxygen, leading to a buildup of lactate as a byproduct.
Lactate dehydrogenase (LDH) (units per liter (U/L) | At baseline and longitudinally at 6 (+/- 14 days) and 12 months (+/- 14 days)
  This parameters has been added to better understand systemic glycolysis in this population in the context of measuring bioenergetics in muscle via fMRS. Normal LDH levels in children vary by age. Normal adult range is 140-280 U/L. An elevated level of lactate dehydrogenase (LDH) in glycolysis indicates an increased rate of anaerobic metabolism.
Trough risdiplam drug levels | At baseline and longitudinally at 6 (+/- 14 days) and 12 months (+/- 14 days)
  Trough risdiplam drug level is measured in nanograms per milliliter from blood samples and indicates the concentration of risdiplam in someone's blood stream. Higher values mean someone has more risdiplam exposure.
  This will only be tested on participants who are taking the drug risdiplam.
Quality of life (QOL) and disability information - Pediatric Quality of Life Inventory (PedsQL) | At baseline and longitudinally at 6 (+/- 14 days) and 12 months (+/- 14 days)
  The Pediatric Quality of Life Inventory (PedsQL) is a 23-item questionnaire measuring health-related quality of life in children and adolescents aged 2-18. Higher scores indicate better quality of life.
QOL and disability information - Pediatric Outcomes Data Collection Instrument (PODCI) | At baseline and longitudinally at 6 (+/- 14 days) and 12 months (+/- 14 days)
  The Pediatric Outcomes Data Collection Instrument (PODCI) is an 83-86 item questionnaire that measures the health-related quality of life for children and adolescents with musculoskeletal disorders aged 2-18. Higher scores indicate better quality of life.
QOL and disability information - SMA Health Index (SMA-HI) | At baseline and longitudinally at 6 (+/- 14 days) and 12 months (+/- 14 days)
  The SMA Health Index (SMA-HI) is a 107 item questionnaire that measures a patient's perception of disease burden in 15 areas of health related to SMA. Higher scores indicate more SMA disease burden

CONTACTS AND LOCATIONS:
Overall Officials: Richard Finkel, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: Description St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols